CLINICAL TRIAL: NCT04669977
Title: Treatment Effects of a Glucoside- and Rutinoside-rich Crude Material in Chemotherapy-induced Peripheral Neuropathy and Related Symptoms
Brief Title: Effects of a Glucoside- and Rutinoside-rich Material in Chemotherapy-induced Peripheral Neuropathy and Related Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N202006058
Record Dates: First submitted 2020-12-09; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Chemotherapy; cyanidin; interleukin; peripheral neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Auxiliary (Experimental): One bottle (600ml/bottle) of sanitized mulberry juice would be sent to participants of the auxiliary group with instructions to consume 50ml of juice diluted with drinking water at room temperature. They are expected to finish the mulberry juice in 10 to 11 days. Measurements of clinical symptoms and blood sampling are conducted on day 1 of every other week for 5 weeks. If clinical measurements or blood extractions fail or miss, a substitute assessment or blood sample will be obtained on day 2 or day 3. The research period for these participants is 29 days (4 weeks). The checkpoints are arranged because patients with oxaliplatin treatment visit the clinic every two weeks, and patients with paclitaxel treatment visit the clinic every week. For patients having docetaxel therapy, the research period is 43 days (6 weeks) because docetaxel is administered every three weeks.
  Interventions: Dietary Supplement: Mulberry juice
- Non-auxiliary (No Intervention): For the non-auxiliary group (control group), patients are informed of their allocation results and they will not consume mulberry juice during the research period but will receive the mulberry juice after the research period.

INTERVENTIONS:
Dietary Supplement: Mulberry juice — One bottle (600ml/bottle) of sanitized mulberry juice would be sent to participants of the auxiliary group with instructions to consume 50ml of juice diluted with drinking water at room temperature. Also, a reminder of the next clinical visit is attached. They are expected to finish the mulberry juice in 10 to 11days instead of 12 days.
  Arms: Auxiliary

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN is common among cancer patients during or after chemotherapy, and the currently available drugs cannot effectively manage the symptoms. Besides, CIPN causes fatigue, anxiety, and depression. CIPN is featured by the interference of interleukin (IL) pathways, among which escalation of IL-17 is predominant, suggesting that IL-17 may be manipulated to reduce the inflammation or the immunological disturbance. Cyanidin, a type of glucosides, has been proved to behave like an IL-17 inhibitor. We have identified a food material that contains large amounts of glucosides and rutinosides - mulberry juice. The current proposal aims to explore the effect of this IL-17 inhibitor-rich material in CIPN and related symptoms. We plan to divide the potential participants into severe pain and mild pain group to conduct two human studies. A single-blinded randomized controlled design is adopted to compare the effects of this crude material between the experimental group and the control group in (1) pain and CIPN of the severe pain participants and (2) fatigue, anxiety, and depression in the mild pain participants. IL and other immune markers will be tested as evidence of improvement of inflammation status. We expect a decrement in pain, CIPN, fatigue, anxiety, and depression severity with the intake of this IL-17 inhibitor-rich material among cancer patients undergoing chemotherapy.

DETAILED DESCRIPTION:
Cancer is at least partially attributable to immunological disturbance, and its treatment causes additional inflammatory problems. Chemotherapy-induced peripheral neuropathy (CIPN), especially that induced by oxaliplatin or Taxanes (including paclitaxel and docetaxel) is common among cancer patients during or after the treatment of chemotherapeutic agents, presented as pain and sensory abnormalities for months, and even persists for years in some patients after the cessation of chemotherapy. Even worse is that currently available drugs cannot effectively manage these conditions. Besides, CIPN causes fatigue, anxiety, and depression, which lower patients' quality of life and determination to fight the disease. Interestingly, CIPN is featured by the interference of interleukin (IL) pathways, among which escalation of IL-17 is predominant, suggesting that IL-17 may be manipulated to reduce the inflammation or the immunological disturbance. Cyanidin, a type of glucosides, has been proved to behave like an IL-17 inhibitor and works in an animal model of skin hyperplasia in reducing the IL-17 levels and severity of hyperplasia. We have identified a food material that contains large amounts of glucosides and rutinosides - mulberry juice. Preliminary findings of an ongoing human study of our team have provided statistical evidence that this crude material effectively relieves clinical symptoms of a disorder associated with inflammation features. The current proposal aims to explore the effect of this IL-17 inhibitor-rich material in CIPN and related symptoms. To avoid confounding effects from pain, we plan to divide the potential participants into severe pain and mild pain group to conduct two human studies. A single-blinded randomized controlled design is adopted to compare the effects of this crude material between the experimental group and the control group in (1) pain and CIPN of the severe pain participants and (2) fatigue, anxiety, and depression in the mild pain participants. IL and other immune markers will be tested as evidence of improvement of inflammation status. We expect a decrement in pain, CIPN, fatigue, anxiety, and depression severity with the intake of this IL-17 inhibitor-rich material among cancer patients undergoing chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible for study 1 (水ffects of mulberry juice on pain and CIPN in participants with severe pain) if they have any cancer and are receiving the oxaliplatin or taxanes (paclitaxel and docetaxel) containing regimen weekly. Other inclusion criteria are (1) age ≥20 and <75 years; (2) performance status (PS) 0-2 according to the Eastern Cooperative Oncology Group (ECOG) scale; (3) life expectancy > 2 months. Visual analog scale (VAS) ≥4. Subjects for study 2 (水ffects of mulberry juice on fatigue, anxiety, and depression in participants with moderate pain) must meet all criteria above with the exception that the VAS should be <4.

Exclusion Criteria:

Patients are excluded if they (1) are not communicable; (2) have received radiotherapy within 4 weeks and cardiac dysfunction due to prior anthracyclines; (3) have symptomatic brain metastasis, symptomatic fluid retention, or severe comorbidities such as uncontrolled diabetes mellitus, severe hypertension or infection; (4) have psychiatric or social conditions that would prevent compliance with treatment, follow-up or adequate informed consent. Pregnant or lactating females are also ineligible.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2020-12-02 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Within 10 weeks
  Pain Assessment
Taiwanese version of Neuropathic pain symptom inventory (NPSI-T) | Within 10 weeks
  To evaluate the detail of pain of the patients, such as the quality of pain, numbness and tingling.
Taiwanese version of the Brief Fatigue Inventory (BFI-T) | Within 10 weeks
  Assessment of the severity of CIPN

SECONDARY OUTCOMES:
Heart rate variability | Within 10 weeks
  Assessment of physiological changes during the research period by using a portable photoplethysmography
General Anxiety Disorder-7 items (GAD-7) | Within 10 weeks
  To measure anxiety levels
Patient Health Questionnaire-9 items (PHQ-9) | Within 10 weeks
  To measure depression levels
Inflammation status | Within 10 weeks
  Evaluated by measuring CRP, known cytokines (IL-6, IL-1β, TNF-α, G-CSF, GM-CSF, and TGF-β), chemokines (IL-8, GRO-α, and MCP-1), and PGE in sera, in addition to the sentinel molecule IL-17A.

CONTACTS AND LOCATIONS:
Overall Officials: El-Wui Loh, PhD, Principal Investigator — Taipei Medical University
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan